CLINICAL TRIAL: NCT06374485
Title: A Phase I, Single-arm, Open-label, Dose-escalation, Safety and Pharmacokinetic Study of AU409 Capsule in Advanced Hepatocellular Carcinoma Patients Who Failed Standard Treatment
Brief Title: Study of AU409 Capsule in Advanced Hepatocellular Carcinoma Patients Who Failed Standard Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU409-LEES-2021-03
Record Dates: First submitted 2024-03-11; First posted 2024-04-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AU409 120mg QD (Experimental): Cohort 1
  Interventions: Drug: AU409
- AU409 210mg QD (Experimental): Cohort 2
  Interventions: Drug: AU409
- AU409 300mg QD (Experimental): Cohort 3
  Interventions: Drug: AU409

INTERVENTIONS:
Drug: AU409 — Oral administration

SUMMARY:
This study is a Phase I, dose-escalation study of AU409 in advanced hepatocellular carcinoma patients who failed standard treatment. A '3+3' dose-escalation design will be utilized to gradually increase the dose of AU409, aiming to assess the safety, tolerability, pharmacokinetics, and preliminary antitumor efficacy of multi-dose AU409 in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 18-75 (inclusive) years of age.
2. Patients with histologically and/or cytologically and/or radiologically confirmed advanced (unresectable or metastatic) hepatocellular carcinoma (HCC) that have failed any of standard treatment (including Immunotherapies and/or Tyrosine Kinase Inhibitor therapies, or Oxaliplatin-based systemic chemotherapies), recurrence, or are intolerant.
3. Before treatment initiation, patients must have previously completed chemotherapy, radiotherapy, interventional therapy for more than 4 weeks (except palliative radiotherapy for bone metastasis). And all treatment-related toxicities (except hair loss, pigmentation, and chemotherapy-related neurotoxicities, etc.) have recovered (≤ level 1 or baseline level).
4. Have at least one evaluable disease lesion based on the modified Response Evaluation Criteria in Solid Tumors (mRECIST).
5. ECOG score of 0 or 1.
6. Patients with Child Pugh class A or some class B (≤7 and no hepatic encephalopathy).
7. Have a life expectancy of >12 weeks.
8. Able to be orally administered.
9. Laboratory examinations must meet the following criteria within 7 days before treatment initiation:

   * Absolute neutrophil count（ANC）≥1.5 × 109/L，platelets（PLT） count ≥75 × 109/L，hemoglobin（HGB）≥90 g/L，and patients are not allowed to receive blood transfusion or other haematopoietic growth factors within 14 days before treatment initiation.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be ≤5.0×upper limit of normal (ULN).
   * Total bilirubin (TBIL) ≤1.5×ULN.
   * Ablumin (ALB) ≥28g/L.
   * Serum creatinine (CRE) ≤1.0×ULN, creatinine clearance rate (CCR) ≥60 mL/min (Cockcroft-Gault equation).
   * International normalized ratio（INR）≤1.5，prothrombin time (PT) ≤1.5×ULN.
10. Have a negative serum pregnancy test for premenopausal women (postmenopausal women who have been menopausal for at least 12 months are considered as infertile). For male patients (including male patients' female spouses of child-bearing potential) and female patients of child-bearing potential must be contraceptive throughout the study and within the 6 months following the last dose of AU409.
11. Patients voluntarily give written informed consent form (ICF).

Exclusion Criteria:

1. Patients of central nervous system metastasis with clinical symptoms (except patients who are asymptomatic, and no disease progression confirmed by MRI diagnosis for more than 28 days).
2. Allergies to any ingredients or excipients in AU409.
3. Treatment with other anticancer therapies (including surgery, radiation therapy, chemotherapy, anti-angiogenic therapy, targeted therapy, or radiofrequency ablation therapy, etc.) or investigational therapy (except patients who stop treatment of Chinese patent medicine or Chinese herbal medicine for more than 7 days, or complete palliative radiotherapy for bone metastasis >2 weeks) within 28 days prior to the first dosing.
4. QTc ≥470 msec during screening period (Fridericia's equation) or with a history of congenital long QT syndrome.
5. Patients with history of gastrointestinal surgery that may change the absorption and activity of drugs in their body (such as total gastrectomy, small bowel resection, external bile shunt, etc.) in combination with refractory hiccups, nausea, vomiting, and other diseases that affect drug absorption (such as peptic ulcer, inflammatory bowel disease, lactose intolerance, malabsorption syndrome or chronic diarrhea, etc.).
6. Patients who require serous effusion for continuous drainage or drug infusion (such as ascites, pleural effusion, etc.), or have undergone portal vein shunt.
7. Patients with gastrointestinal perforation and/or fistula, abdominal abscess, visceral fistula, intestinal obstruction, hepatic encephalopathy, portal vein and inferior vena cava cancer thrombus within 3 months prior to the treatment initiation.
8. Patients have gastrointestinal bleeding (including esophageal or gastric varices, local active ulcer lesions, etc.), or have a clear bleeding tendency, or are receiving anticoagulation/thrombolytic therapy within 3 months before treatment initiation. Positive result of occult blood needs to identifythe causes.
9. Patients with interstitial lung disease, non-infectious pneumonia.
10. History of allogeneic stem cell transplantation or organ transplantation.
11. Patients who receive major surgery (except biopsy and puncture) or with major trauma within 28 days before treatment initiation.
12. Patients with infectious diseases that affect daily activities or require systemic treatment (such as the use of hormones, antibiotics, antifungal drugs, antiviral drugs, and oxygen inhalation), including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.
13. Uncontrolled diseases, including a) New York Heart Association (NYHA) Class II or higher heart failure, b) Severe/unstable angina pectoris, c) Primary cardiomyopathy, d) Myocardial infarction or coronary/peripheral artery bypass surgery occurred within 6 months before treatment initiation, e) Uncontrollable high blood pressure, f) Severe arrhythmia requiring medication or intervention, g) Echocardiographic left ventricular ejection fraction <50% during the screening period, h) Deep vein thrombosis/arterial thrombosis /Pulmonary vein embolism occurred within 2 months before treatment initiation, i) Cerebrovascular accident or transient ischemic attack occurred within 6 months before treatment initiation, j) Ocular lens disease (such as cataract), k) Diabetes that has not been effectively controlled, l) Thyroid diseases that have not been effectively controlled, m) Urine protein≥2+ and quantity of 24-hour urine protein ≥1.0g.
14. Human immunodeficiency virus infection (HIV 1/2 antibody positive).
15. HBV infection (HBsAg positive and HBV DNA ≥2000 IU/mL); Hepatitis C virus (HCV) antibody is positive and HCV RNA>103 copies/ml; HBsAg and HCV antibodies are both positive.
16. Patients with tuberculosis (TB) who need to receive/are receiving anti-TB treatment within 1 year before treatment initiation.
17. Pregnant or nursing；
18. Patients complicated with other malignant tumors within 5 years before treatment initiation, except various in situ tumors, skin basal cell carcinoma or squamous cell carcinoma that have been cured in the past, local prostate cancer receiving radical operation, and in situ breast ductal carcinoma receiving radical operation.
19. Patients with other severe, acute, chronic, or psychiatric illnesses that may increase the risk of treatment or may interfere with interpretation of the trial results. And patients with alcoholism, smoking addiction, drug abuse, and other circumstances that are not conductive to the treatment or explain adverse events, thereby contributing to decrease study compliance.
20. Other conditions that are not suitable for participating in the study in the opinion of investigator.
21. Patients who were treated with pentamidine prior to treatment initiation or during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | At the end of Cycle 1 (each cycle is 28 days)
  To determine the maximum tolerated dose (MTD) and the recommended phase II dose (R2PD).

SECONDARY OUTCOMES:
Maximum Tolerated Dose | Through study completion, an average of 2 years
  If 2 or more out of 3 or 6 patients at a dose level develop DLTs, the dose will be considered as "intolerable dose", and the preceding dose level is defined as the Maximum Tolerated Dose (MTD).
Recommended Phase 2 Dose | Through study completion, an average of 2 years
  RP2D will be determined in accordance with occurrence of the DLTs and AEs.
Objective Response Rate | Through study completion, an average of 2 years
  The proportion of patients whose best efficacy is CR and PR observed throughout the study from enrollment to disease progression.
Disease Control Rate | Through study completion, an average of 2 years
  The proportion of patients whose best efficacy is CR, PR, and SD throughout the study from enrollment to disease progression.
Duration of Response | Through study completion, an average of 2 years
  The time from the first tumor evaluation as CR or PR to the first evaluation as PD or death from any cause during the study.
Progression-free Survival | Through study completion, an average of 2 years
  The time from enrollment until the disease progression or death from any cause.
Overall Survival | Through study completion, an average of 2 years
  The time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No